CLINICAL TRIAL: NCT05601440
Title: A Liquid-biopsy Informed Platform Trial to Evaluate Treatment in CDK4/6-inhibitor Resistant ER+/HER2- Metastatic Breast Cancer
Brief Title: Liquid-biopsy Informed Platform Trial to Evaluate CDK4/6-inhibitor Resistant ER+/HER2- Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I241
Record Dates: First submitted 2022-10-25; First posted 2022-11-01 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Observation; niraparib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Substudy A - Monitoring (Experimental)
  Interventions: Other: Observation
- Substudy B - RP-6306 + Gemcitabine - Arm Permanently Closed (Experimental)
  Interventions: Drug: RP-6306; Drug: Gemcitabine
- Substudy C - Niraparib + Fulvestrant (Experimental)
  Interventions: Drug: Niraparib; Drug: Fulvestrant
- Substudy D - RP-6306 + RP-3500 - Arm Permanently Closed (Experimental)
  Interventions: Drug: RP-6306; Drug: RP-3500

INTERVENTIONS:
Drug: RP-6306 — Dose and schedule will be assigned at enrolment
  Other Names: Lunresertib
  Arms: Substudy B - RP-6306 + Gemcitabine - Arm Permanently Closed; Substudy D - RP-6306 + RP-3500 - Arm Permanently Closed
Drug: Gemcitabine — Dose and schedule will be assigned at enrolment
  Arms: Substudy B - RP-6306 + Gemcitabine - Arm Permanently Closed
Other: Observation — Monitoring arm
  Arms: Substudy A - Monitoring
Drug: Niraparib — Dose and schedule will be assigned at enrolment
  Arms: Substudy C - Niraparib + Fulvestrant
Drug: Fulvestrant — Dose and schedule will be assigned at enrolment
  Arms: Substudy C - Niraparib + Fulvestrant
Drug: RP-3500 — Dose and schedule will be assigned at enrolment
  Other Names: Camonsertib
  Arms: Substudy D - RP-6306 + RP-3500 - Arm Permanently Closed

SUMMARY:
This study is being done to answer the following question: Can testing breast cancer for DNA abnormalities or "biomarkers" help predict which patients are most likely to be helped by certain treatments? The pre-study screening is being done to test a sample of blood (or tumour tissue) for biomarkers to see if patients can participate in the study

DETAILED DESCRIPTION:
This is a 2-stage master protocol with multiple substudies testing investigational drugs/drug combinations in patients with CDK4/6-inhibitor resistant ER+/HER2- metastatic breast cancer. First line endocrine therapy (1LET, aromatase inhibitors; AI) improve clinical outcomes, but are not curative, and acquired resistance develops (median ~2 years). CDK4/6i-resistant MBC is a clinical unmet need, and is marked by numerous potential resistance alterations / mechanisms. Currently, most patients receive second line (2L) ET (e.g., fulvestrant) which has a median progression-free survival (PFS) of ~2 months in this setting. Circulating tumour DNA (ctDNA) and circulating tumour cells (CTCs) are detectable in peripheral blood in >90% of patients with MBC.

Patients who wish to participate but progression has not yet occurred may be enrolled in the monitoring substudy and followed until progression. This monitoring component of IND.241 aims to characterize the molecular and clinical features of CDK4/6i resistance as it occurs after first line CDK4/6i + AI. Besides addressing the principal objectives described above (ctDNA genotyping and evaluation of dynamic changes in ctDNA and CTC levels), banked samples will create a biorepository for interrogation of emerging assays (e.g., DNA methylation, CTC protein or single cell analyses) that may have prognostic or predictive application. These data will inform future efforts that may consider intervention prior to clinical treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically and/or cytologically confirmed, advanced / metastatic breast cancer, ER >10% and not HER2 overexpressing/amplified as per ASCO/CAP criteria. Patients with locally advanced or inflammatory disease without distant metastases that is potentially resectable or treatable with curative intent are not eligible
* All patients must have a formalin fixed paraffin embedded tissue block (from primary or metastatic tumour) available and must have provided informed consent for the release of the block
* Patients must have had objective disease progression demonstrated on (defined as while taking or within 8 weeks of the last dose) first line CDK4/6i + ET for MBC. Patients who discontinued CDK4/6i + ET without disease progression more than 8 weeks prior to objective disease progression (toxicity, patient request) are not eligible. Patients must have received at least 24 weeks of first line CDK4/6i + ET therapy
* Presence of clinically and/or radiologically documented disease. All radiology studies must be performed within 21 days prior to enrollment (within 28 days if negative). All patients must have measurable disease as defined by RECIST 1.1.
* The criteria for defining measurable disease are as follows:

  * Chest x-ray ≥ 20 mm
  * CT scan (with slice thickness of 5 mm) ≥ 10 mm: longest diameter
  * Physical exam (using calipers) ≥ 10 mm
  * Lymph nodes by CT scan ≥ 15 mm: measured in short axis
* Patients must be ≥ 18 years of age
* Patients must have an ECOG performance status 0 or 1
* Patients must have a life expectancy ≥ 3 months.
* Hemoglobin ≥90 g/L*
* Absolute neutrophils ≥ 1.5 x 10^9/L (1500/µL)
* Platelets ≥ 100 x 109/L (100 x 10^3/µL)
* Bilirubin ≤ 1.5 x ULN (upper limit of normal)**
* AST & ALT ≤ 2.5 x ULN
* ≤ 5.0 x ULN if patient has liver metastases
* Serum creatinine ≤ 1.5 x ULN, Creatinine clearance ≥50 mL/min
* All patients must have received at least 24 weeks of prior CDK4/6i in combination with first line ET for advanced or metastatic disease and have had disease progression on or within 8 weeks of the last dose of CDK4/6i. Patients who have progressed on, or within 12 months of completion of adjuvant therapy with an aromatase inhibitor may be treated with fulvestrant instead of an aromatase inhibitor combined with CDK4/6 inhibitor.

In addition, the following systemic therapies may have been given after CDK4/6i / ET prior to screening / enrollment to this study:

* For enrollment to "second line" substudies:

  - An additional single agent non-fulvestrant/SERD endocrine therapy in the palliative setting is permitted provided patient remains eligible for and can access fulvestrant treatment. Patients who have received prior fulvestrant/SERD are not eligible for fulvestrant containing substudies. Contact CCTG in case of any other prior endocrine therapy other than an aromatase inhibitor or tamoxifen.
* For enrollment to "third line" substudies:

  * Non-SERD endocrine therapy and targeted agents alone or in combination.
  * Patients who have received a prior targeted agent may not be eligible for substudies that contain the same class of agent. Contact CCTG.
  * Note: if a patient has not had fulvrestrant/SERD prior to enrollment to "3rd line: substudy, single agent fulvestrant/SERD must be given prior to enrollment (unless not possible for reasons such as fulvestrant/SERD not standard of care / not funded in province, patient cannot receive intramuscular injection; contact CCTG for other scenarios).
* Patients may also have received adjuvant/neoadjuvant systemic therapies; however cytotoxic chemotherapy or antibody drug conjugates (ADC) in the palliative setting are not permissible.
* Patients receiving LHRH agonists (for example premenopausal patients) may continue, but may not start LHRH agonist within 12 weeks of enrollment.
* Consult CCTG for other scenarios (for example where short course of other ET is given prior to CDKi + ET, patients who have received investigational drugs, vaccines or immunotherapies) as certain patients may be eligible.
* All reversible prior toxicity related to prior therapies must have recovered to grade ≤ 1 (consult CCTG in the case of irreversible toxicity) and have adequate washout as follows (screening may occur during the washout period): Longest of the following (for questions or any proposed variance, please discuss with CCTG prior to patient enrollment): Two weeks; 5 half-lives for investigational agents; standard cycle length of standard therapies
* Patients must not have received a transfusion (platelets or red blood cells) or colony stimulating factors ≤ 4 weeks prior to initiating treatment substudy therapy.
* Surgery: Prior surgery is permitted provided that a minimum of at least 28 days have elapsed between any major surgical procedure and date of enrollment, and that wound healing has occurred.
* Radiation: Prior external beam radiation is permitted provided a minimum of 28 days (4 weeks) have elapsed between the last dose of radiation and date of enrollment. Exceptions may be made for low-dose, non-myelosuppressive radiotherapy after consultation with CCTG. Concurrent radiotherapy is not permitted.
* Patients must be registered and provide consent prior to blood collection for screening. The screening blood sample cannot be sent for analysis prior to screening registration.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to both screening registration as well as enrollment to a specific substudy to document their willingness to participate.
* Patients must be accessible for treatment and follow up. Patients enrolled on this trial must be treated and followed at the participating centre
* In accordance with CCTG policy, substudy treatment is to begin within 2 working days of patient enrollment.
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method.

Exclusion Criteria:

* Patients with a history of other malignancies, including Myelodysplastic syndrome (MDS) or Acute myeloid leukemia (AML) except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other malignancies curatively treated with no evidence of disease for ˃ 2 years and which do not require ongoing treatment.
* Patients with active or uncontrolled infections or with serious illnesses or medical conditions which would not permit the patient to be managed according to protocol.

  * Infection includes but is not limited to active infection requiring systemic therapy and active or known human immunodeficiency virus (HIV) with detectable viral load, known hepatitis B surface antigen or positive hepatitis C antibody
  * Pneumonitis or any history of pneumonitis requiring steroids (any dose)
  * Participant has received a live vaccine within 30 days of planned start of study therapy. COVID19 vaccines that do not contain live viruses are allowed.
  * Known primary immunodeficiency
* Patients with recent clinically significant cardiac disease, including:

  * angina pectoris, symptomatic pericarditis, coronary artery bypass grafting, coronary angioplasty, or stenting, or myocardial infarction in the previous 12 months;
  * history of documented congestive heart failure (New York Heart Association functional classification III-IV) or cardiomyopathy
  * uncontrolled hypertension (per Canadian guidelines)
* All patients should have a LVEF ≥ 50%.
* Patients with HER2 positive breast cancer (based on the most recent assessment, according to ASCO/CAP criteria).
* History of hypersensitivity to any of the study drugs or their components.
* Patients may not receive concurrent treatment with other anti-cancer therapy (other than bone-targeted therapy, if already taking and stable) or investigational agents while on protocol therapy.
* Patients with prior allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
* Pregnant or breastfeeding women.
* Patients with history of central nervous system metastases or spinal cord compression unless they have received definitive treatment such as resection or radiation, are clinically stable and do not require corticosteroids; corticosteroids must have been discontinued at least 7 days prior to enrollment.
* Patients who are unable to swallow oral medication and/or have impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g. Crohn's disease, ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, active bowel inflammation (e.g. diverticulitis) or small bowel resection), unless agreed with CCTG (exceptions may be given if a parenteral treatment substudy is available/appropriate).
* Patients with a history of non-compliance to medical regimens.
* See Section 7.3 and individual treatment substudies for a list of concomitant medications that are not permitted.
* Many substudies include drugs that have a risk for thrombocytopenia; therefore, participants should be advised to use caution when taking oral anticoagulants (e.g. warfarin) and antiplatelet drugs (e.g. aspirin).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 484 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate whether biomarker selection improves outcomes as assessed by RECIST 1.1 for overall response rate | 5 years
Evaluate whether biomarker selection improves outcomes as assessed by RECIST 1.1 for clinical benefit rate | 5 years

SECONDARY OUTCOMES:
Number and severity of adverse events | 5 years
Progression-free survival (PFS) | 5 years
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: David Cescon, Study Chair — University Health Network, Princess Margaret Hospital, Toronto ON Canada; John Hilton, Study Chair — Ottawa Hospital Research Institute; Nathalie Levasseur, Study Chair — BCCA - Vancouver Cancer Centre; Stephen Chia, Study Chair — BCCA - Vancouver Cancer Centre; Moira Rushton, Study Chair — Ottawa Hospital Research Institute
Locations (10):
- Canada (10):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - BCCA - Kelowna, Kelowna, British Columbia
  - BCCA - Vancouver, Vancouver, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - The Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No